CLINICAL TRIAL: NCT06601517
Title: A Phase I, Open-Label, Single-Arm, Fixed-Sequence Study to Evaluate the Effect of Repeated Administration of HDM1002 on the Pharmacokinetics of Repaglinide, Atorvastatin, Digoxin and Rosuvastatin in Healthy and Overweight Adult Chinese Subjects
Brief Title: A Drug-Drug Interaction (DDI) Study of HDM1002 With Repaglinide, Atorvastatin, Digoxin and Rosuvastatin in Healthy Subjects and Overweight Subjects.
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Hangzhou Zhongmei Huadong Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HDM1002-106
Record Dates: First submitted 2024-09-03; First posted 2024-09-19 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Healthy Adult Subject; Overweight Subject
Keywords: HDM1002; Glucagon-Like Peptide-1 Receptor Agonists
MeSH Terms: interventions — repaglinide; Atorvastatin; Digoxin; Rosuvastatin Calcium

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- HDM1002 with Repaglinide, Atorvastatin, Digoxin and Rosuvastatin (Experimental): Period 1: Single dose of repaglinide, atorvastatin, digoxin and rosuvastatin
  Period 2: Once daily dose of HDM1002
  Period 3: Single dose of repaglinide, atorvastatin, digoxin and rosuvastatin with once daily dose of HDM1002
  Interventions: Drug: Repaglinide; Drug: Atorvastatin; Drug: Digoxin; Drug: Rosuvastatin; Drug: HDM1002

INTERVENTIONS:
Drug: Repaglinide — Single dose; Administered orally
Drug: Atorvastatin — Single dose; Administered orally
Drug: Digoxin — Single dose; Administered orally
Drug: Rosuvastatin — Single dose; Administered orally
Drug: HDM1002 — Administered orally

SUMMARY:
The purpose of this study is to characterize the effect of HDM1002 on the PK of single dose of repaglinide, atorvastatin, digoxin and rosuvastatin in healthy adult subjects. The safety and tolerability of HDM1002 with repaglinide, atorvastatin, digoxin and rosuvastatin when given separately or together will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. According to the medical history, clinical laboratory test results, vital sign measurements, 12 lead ECG results, and physical examination results during the screening period, the investigator considers the subject to be in good general health.
2. Age range of 18-45 years old (including range), no limit to gender.
3. Male subject weighed ≥50.0 kg, female subject weighed ≥45.0 kg, and a body mass index (BMI) within the range of 19.0 - 30.0 kg/m2 (including cut-off values).

Exclusion Criteria:

1. Subject has a history or family history of medullary thyroid cancer, thyroid C-cell hyperplasia, or multiple endocrine neoplasia type 2 (MEN2), or calcitonin≥50 ng/L during the screening period.
2. History of chronic pancreatitis or an episode of acute pancreatitis within 3 months prior to screening.
3. History of acute cholecystitis attack within 3 months prior to screening.
4. Subject judged by investigator has dysphagia, diseases or conditions that affect gastric emptying, or affect the absorption of gastrointestinal nutrients, such as bariatric surgery or other gastrectomy, irritable bowel syndrome, dyspepsia, etc.
5. History of previous surgery that will affect the absorption, distribution, metabolism, and excretion of drugs or plan to undergo surgery during the study period.
6. During screening period, any abnormalities in physical examination, electrocardiogram, laboratory tests, and vital signs which are of clinically significant .
7. Taken or planned to take any drug that effect liver enzyme or transporter activity within 28 days prior to taking the investigational drug.
8. History of clinically significant cardiovascular and cerebrovascular disease within 6 months prior to screening or at the time of admission.
9. Presence of clinically significant ECG results judged by the investigator at screening.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2025-02 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
AUC[0-∞] | Period 1 and Period 3: Day 1-Day 16
  Pharmacokinetics (PK) parameter of repaglinide, atorvastatin, digoxin and rosuvastatin: Area under the curve from time 0 hour to ∞
AUC[0-t] | Period 1 and Period 3: Day 1-Day 16
  PK parameter of repaglinide, atorvastatin, digoxin and rosuvastatin: Area under the curve from time 0 to t hour
Cmax | Period 1 and Period 3: Day 1-Day 16
  PK parameter of repaglinide, atorvastatin, digoxin and rosuvastatin: Maximum observed concentration

SECONDARY OUTCOMES:
Tmax | Period 1 and Period 3: Day 1-Day 16
  PK parameter of repaglinide, atorvastatin, digoxin and rosuvastatin: Time to maximum plasma concentration
t1/2 | Period 1 and Period 3: Day 1-Day 16
  PK parameter of repaglinide, atorvastatin, digoxin and rosuvastatin: Half life
CL/F | Period 1 and Period 3: Day 1-Day 16
  PK parameter of repaglinide, atorvastatin, digoxin and rosuvastatin: Apparent Clearance
Vz/F | Period 1 and Period 3: Day 1-Day 16
  PK parameter of repaglinide, atorvastatin, digoxin and rosuvastatin: Apparent volume of distribution
Adverse events (AEs) | Period 1 and Period 3: Day 1-Day 16, Period 2: Day 1-Day 35
  Number of subjects reporting AEs

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, China